CLINICAL TRIAL: NCT01442740
Title: 15-Degree Reverse Trendelenburg Position for FESS
Brief Title: 15-Degree Tilt, Head Up, Feet Down Body Position for Sinus Surgery Patients
Acronym: RTP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Amin Javer, Principal Investigator, St. Paul's Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RTP-2011
Record Dates: First submitted 2011-09-26; First posted 2011-09-28 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Sinusitis
Keywords: Functional Endoscopic Sinus Surgery; Reverse Trendelenburg Position
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 15-degree Reverse Trendelenburg Position (Experimental): Patients will be placed on the operating table in a position where the lower extremities are leveled lower than the head and neck. The angle of incline will be set at 15 degrees from the horizontal.
  Interventions: Procedure: Reverse Trendelenburg Position
- 0-degree Supine Position (No Intervention): Patients will be placed on the operating table in the standard, 0-degree supine position.

INTERVENTIONS:
Procedure: Reverse Trendelenburg Position — Patients will be placed on the operating table in a head up, feet down, tilt position (15 degree tilt to the horizontal). This is in contrast to the standard of care, 0-degree supine position.
  Other Names: RTP
  Arms: 15-degree Reverse Trendelenburg Position

SUMMARY:
Functional Endoscopic Sinus Surgery (FESS) is normally performed in our centre in a 0-degree supine position, with the patient laying flat. This study will be investigating whether changing patients to a 15-degree head up, feet down position will improve field of view and reduce blood loss during surgery. The 15-degree head up, feet down position has been used in other circumstances, such as brain surgery and for severely obese patients where airways can be blocked due to lying flat. Every 15 minutes, blood pressure, heart rate and field of view according to the Boezaart nasal scope scaling system will be recorded.

DETAILED DESCRIPTION:
Our objective is to determine whether 15-degree RTP during FESS will influence intra-operative blood loss and surgical field scores when compared to patients in a supine position.

Our hypothesis is that the 15-degree RTP position is not inferior to the supine position in reducing intra-operative blood loss and improving surgical field view during FESS.

Specific Aims

Aim 1: To determine the effect of 15-degree RTP on total blood loss, time of surgery and endoscopic surgical view, when compared with patients in the supine position, during FESS.

Participants will have their sinus cavities assessed by rigid endoscopy during surgery. The Boezaart scaling system will be used as our primary endoscopic surgical field measure. Total Blood Loss (TBL), Mean Arterial Pressure (MAP), pulse rate and Time of Surgery (TOS) will be recorded intra-operatively by the anesthesiologist and supporting nurse staff. The results of this experiment will determine whether utilizing the 15-degree RTP is effective to reduce blood loss during ESS.

Background and significance:

Chronic Rhinosinusitis (CRS) is associated with nasal obstruction, discolored nasal discharge, facial congestion or pressure that lasts at least twelve weeks (1,2). Nasal polyposis may also be present with CRS (1,2). Corticosteroids and medicated nasal irrigations are recommended as preliminary treatment options3. Sinus surgery is recommended for patients whose symptoms are refractory to maximal medical management. FESS has evolved to become the preferred surgical method for treating CRS and other sinus related diseases4. When compared to the previous open craniofacial approach, this technique has been found to be less invasive, low-risk and reduces operating time with improved post-operative outcomes4. FESS performed in the supine position has been the standard at the St. Paul's Sinus Centre. Surgeon experience has indicated that patients in a 0-degree operating position, allows for consistent orientation of the sinus anatomy. However, bleeding within the surgical area can obscure endoscopic field of view, increasing risk for surgical complications which may include cerebrospinal fluid leak, hemorrhage, infection and damage to the optic nerve and internal carotid artery (4,6). There are several factors available to control hypotension during surgery such as the use of total intravenous anesthesia (TIVA), pre-operative topical treatment with steroids, local vasoconstrictors and patient position4.

TIVA has been observed to reduce intra-operative hemorrhage by lowering mean arterial pressure (MAP) when compared to inhalational anesthesia during ESS5. The use of corticosteroids prior to surgery has been found to reduce peri-operative blood loss (6). Results indicate that TIVA and pre-operative steroid treatment can significantly lower surgical grade scores by improving endoscopic visualization (5,6). However, altering patient position during the operation may provide a simple option to further reduce the presence of blood within the surgical field.

The Reverse Trendelenburg Position (RTP) is a head-up, feet-down tilt varying from 10 to 30 degrees (7). When used in surgery, RTP has been found to reduce hydrostatic forces and venous congestion (6,7). In morbidly obese patients where anesthesia can alter respiratory function RTP has been identified as a safe intra-operative procedure, improving oxygenation with minimal MAP changes (9). This position has been found to reduce intra-cranial pressure during craniotomy and thereby, decreasing surgical risks for cerebral swelling and herniation (8).

The role of RTP and other factors related to intra-operative blood loss during FESS has recently been examined. Ko et al. (2008) equally randomized 60 CRS patients to receive FESS while in the 10-degree RTP or complete supine position. Patients with CRS with or without nasal polyposis, mild or moderate hypertension, diabetes, chronic renal disease, and other uncritical medical conditions were included in the study (10). Patients were excluded if they had severe or uncontrolled cases of hypertension, cardiovascular disease and preoperative use of anticoagulant medication (10). All patients received a combination of intravenous and inhaled anesthesia. This was induced with fentanyl, xylocaine, propofol and cisatracurim. Desflurane or sevoflurane were used intra-operatively to maintain anesthesia (10). In addition, a 1% solution of lidocaine hydrochloride, a local anesthetic, and adrenaline at a dilution of 1:80,000 was injected into the surgical field and pterygopalatine fossa. Total blood loss (TBL) was measured from the suction bottle during the surgery by an OR nurse. Blood loss per minute (BL/Min) was calculated from dividing the TBL by the total time of the surgery. The Boezaart grading system was used to evaluate the effect of bleeding within the surgical field (SF). The inverse trendelenburg position was found to significantly reduce TBL (P < 0.001), BL/Min (P < 0.001) and SF score (P < 0.004).

Due to the highly vascularized nature of the paranasal sinuses, small amounts of blood can cause substantial impairment to endoscopic view. The RTP reduces venous return and cardiac output by retaining blood in the lower parts of the body (10,11). As a result, reduced intraoperative blood loss has been reported in previous studies employing this operating position during surgery (10,11,12). Although RTP has been utilized in Otorhinolaryngology, the previously mentioned study used a combination of total intravenous and inhaled anesthesia for study subjects (10). Previous literature has shown that TIVA can reduce intra-operative blood loss when compared to inhaled anesthesia5. We aim to evaluate if 15-degree RTP with patients receiving TIVA and preoperative steroid treatment can reduce endoscopic visual impairment.

Experimental Design and Methods:

Research Method:

Randomized unblinded, prospective study

Recruitment of CRS patients

Patients requiring endoscopic sinus surgery will be approached to partake in this study. These patients are individuals who have failed conventional medical therapy and require the expertise of a tertiary rhinologist in treating their sinus disease. This tertiary based rhinology centre averages 6000 outpatient visits and >400 FESS cases a year. This is the busiest rhinology centre in Western Canada. The site coordinator or one of the Principal Investigator's designates will describe the study design to the patients. Patients will have up to one month prior to surgery to sign the consent form if they plan to partake in the study. Patients placed in the study will be provided with the direct line to the St. Paul's Sinus Centre and therefore can talk to any of the co-investigators if they have any questions or concerns.

Inclusion Criteria:

* Patients 19 years of age or older
* Patients who will undergo primary or revision functional endoscopic sinus surgery (FESS)
* Patients with CRS with or without polyposis

Exclusion Criteria:

* Patients under the age of 19
* Patients with a history of coagulation disorders
* Patients with severe or uncontrolled cases of hypertension and cardiovascular disease
* Patients undergoing sinonasal tumor resection

Experimental and Control Arm All patients are treated with a one-week course of prednisone 20mg once a day and oral antibiotics (clavulin or clindamycin if penicillin allergic) prior to surgical intervention. Patients will be randomized to the experimental (15-degree RTP) or control (supine) arm based on a closed envelope system.

Procedure

Pre-Operative:

* Obtain informed consent of 64 patients prior to surgery
* Randomize patients to the experimental (15-degree RTP) arm or the control (supine position) arm.
* 32 patients will receive FESS while in the 15-degree RTP position
* 32 patients will receive FESS while in the standard supine (0-degree) position
* Pre-existing health conditions, current medication and patient demographics (age, sex) will be recorded
* Patients will be instructed to take the standard pre-operative medications used at St. Paul's Hospital (prednisone and antibiotics for 1 week).

Intra-operative:

* Patients will initially be placed in a 0-degree supine position, where blood pressure and pulse rate will be recorded.
* All patients will undergo total intravenous anesthesia, with a prescribed infusion administered by the residing anesthetist. Anesthesia infusions will be documented and recorded.
* The Principal Investigator or one of his designates will electronically calibrate the operating table to bring patients in the experimental arm of the study to the 15-degree RTP. Those in the control arm will remain in the supine position.
* Primary Outcome Measures:

  * MAP, pulse rate and endoscopic field view will be recorded every 15 minutes intra-operatively.
  * Once the procedure is complete, total time of surgery and total estimated blood loss will be recorded.
  * Blood loss per minute will be calculated using total blood loss divided by total operating time.

Aim 1: To determine the effect of 15-degree RTP on total blood loss, time of surgery and endoscopic surgical field view when compared with patients in the supine position, during FESS.

Primary outcome measures will be documented at periodic intervals intra-operatively and at the completion of surgery. The Principal Investigator or one of his designates will record MAP, pulse rate and endoscopic surgical field score every 15 minutes from the start of surgery. Documentation of MAP, pulse rate, and endoscopic surgical field score at periodic intervals is not standard practice during surgery and it will only be done on study patient cases. Once the procedure is completed, total blood loss and time of surgery will be recorded. The total amount of blood lost will be calculated from the suction bottle and measured in milliliters after surgery. This will be confirmed by the circulating nurse and the anesthetist. Total time of surgery will be recorded in minutes, by the circulating nurse and the anesthetist. In certain circumstances the operation may be extended due to unexpected complications, therefore total blood loss may increase due to prolonged surgery. To determine blood loss per minute (mL/min), total estimated blood loss will be divided by time of surgery. Ko et al (2008) previously calculated blood loss per minute with the above formula in their analysis of the role of RTP during endoscopic sinus surgery.

The Boezaart intra-operative surgical field scale will be used to grade the level of bleeding during surgery. This 0 to 5-point scale will be used to outline the amount of suction required to rid the area of blood disrupting vision. A score of 0 is given for an area with no bleeding, 1 for slight bleeding with no suction required, 2 for slight bleeding requiring suction, 3 for moderate bleeding which improves for several seconds once suction has occurred, 4 for moderate bleeding which restarts directly after suctioning and 5 for severe bleeding which occurs faster then can be removed (12).

Data Collection and Statistical Analysis

Discussion with a statistician indicated that based on a previous study10, a population size of 64 patients would be needed to achieve a power rating of 80%. Both the experimental and control arms each will have 32 patients enrolled. To determine the sample size, a confidence interval of 95% was utilized to create a responsive range of double the standard deviation. In consideration of the location and vascularity of the paranasal sinuses, a Boezaart score of 3 is expected during surgery. Clinically significant change in intra-operative bleeding will be defined as a change in Boezaart scoring by 20%, or one point in relation to the scale. All data collected for this study will be gathered in a password protected Microsoft Excel spreadsheet file. Each patient will be assigned unique identification allowing for no patient data to be recorded. The Microsoft Excel database will include:

* Age
* Sex
* Pre-existing health conditions
* Current medications
* Lund-Kennedy CT score
* CRS with or without polyposis
* Primary or revision surgery
* Anesthesia infusion
* Surgical position (15-degree RTP or Supine)
* MAP (15 minute intervals)
* Pulse rate (15 minute intervals)
* Endoscopic surgical field scores (15 minute intervals)
* Intra-operative complications
* Microdebrider usage
* Total blood loss
* Total time of surgery

Risks No adverse risks are expected from placing patients in the experimental 15-degree reverse trendelenburg position. Patient care will not be compromised at any time during surgery. Patients will be able to withdraw from the study at any stage without affecting the quality of the medical care they receive.

Difficulties and Limitations

Aim 1: No difficulties are expected. Standard practice during FESS at the St. Paul's Sinus Centre is to document total time of surgery and blood loss on anesthetist and nurse progress notes, and post-operative surgical reports. For best results, we have included periodic measurement of MAP, pulse rate and endoscopic surgical field view at 15-minute intervals intra-operatively. Unexpected or sudden adverse events during surgery may hinder periodic assessment of our primary outcome measures, as priority will be given to patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo primary or revision functional endoscopic sinus surgery (FESS)
* Patients with CRS with or without nasal polyposis

Exclusion Criteria:

* Patients with a history of coagulation disorders
* Patients with severe or uncontrolled cases of hypertension and cardiovascular disease
* Patients undergoing sinonasal tumor resection

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Boezaart intra-operative surgical field scale | Every 15 minutes for the duration of the surgery
  The Boezaart intra-operative surgical field scale will be used to grade the level of bleeding during surgery. This 0 to 5-point scale will be used to outline the amount of suction required to rid the area of blood disrupting vision. A score of 0 is given for an area with no bleeding, 1 for slight bleeding with no suction required, 2 for slight bleeding requiring suction, 3 for moderate bleeding which improves for several seconds once suction has occurred, 4 for moderate bleeding which restarts directly after suctioning and 5 for severe bleeding which occurs faster then can be removed

SECONDARY OUTCOMES:
Intra-operative vital signs | Every 15 minutes for the duration of surgery.
  The Principal Investigator or one of his designates will record mean arterial pressure, pulse rate and endoscopic surgical field score (5 point system describing clarity of surgical field of view) every 15 minutes from the start of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Amin R Javer, MD, FRCSC, FARS, Principal Investigator — St. Paul's Hospital
Locations (1):
- E.N.T. Clinic, St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Rosenfeld RM. Clinical practice guideline on adult sinusitis. Otolaryngol Head Neck Surg. 2007 Sep;137(3):365-77. doi: 10.1016/j.otohns.2007.07.021. PMID 17765760
- [Background] Meltzer EO, Hamilos DL. Rhinosinusitis diagnosis and management for the clinician: a synopsis of recent consensus guidelines. Mayo Clin Proc. 2011 May;86(5):427-43. doi: 10.4065/mcp.2010.0392. Epub 2011 Apr 13. PMID 21490181
- [Background] Desrosiers M, Hussain A, Frenkiel S, Kilty S, Marsan J, Witterick I, Wright E. Intranasal corticosteroid use is associated with lower rates of bacterial recovery in chronic rhinosinusitis. Otolaryngol Head Neck Surg. 2007 Apr;136(4):605-9. doi: 10.1016/j.otohns.2006.10.028. PMID 17418259
- [Background] Albu S, Gocea A, Mitre I. Preoperative treatment with topical corticoids and bleeding during primary endoscopic sinus surgery. Otolaryngol Head Neck Surg. 2010 Oct;143(4):573-8. doi: 10.1016/j.otohns.2010.06.921. PMID 20869570
- [Background] Wormald PJ, van Renen G, Perks J, Jones JA, Langton-Hewer CD. The effect of the total intravenous anesthesia compared with inhalational anesthesia on the surgical field during endoscopic sinus surgery. Am J Rhinol. 2005 Sep-Oct;19(5):514-20. PMID 16270608
- [Background] Nair S, Collins M, Hung P, Rees G, Close D, Wormald PJ. The effect of beta-blocker premedication on the surgical field during endoscopic sinus surgery. Laryngoscope. 2004 Jun;114(6):1042-6. doi: 10.1097/00005537-200406000-00016. PMID 15179210
- [Background] SHANE SM, ASHMAN H. The prevention of postoperative shock and postanesthesia hypotension by use of the reverse Trendelenburg position during surgery under light, etherless, general anesthesia. Am J Surg. 1957 Jul;94(1):102-7. doi: 10.1016/0002-9610(57)90626-8. No abstract available. PMID 13424879
- [Background] Rolighed Larsen JK, Haure P, Cold GE. Reverse Trendelenburg position reduces intracranial pressure during craniotomy. J Neurosurg Anesthesiol. 2002 Jan;14(1):16-21. doi: 10.1097/00008506-200201000-00004. PMID 11773818